CLINICAL TRIAL: NCT01737528
Title: Society of Thoracic Surgeons and American College of Cardiology Transcatheter Valve Therapy Registry (STS/ACC TVT Registry).
Brief Title: STS/ACC Transcatheter Valve Therapy Registry (TVT Registry)
Acronym: TVTR
Status: Recruiting | Type: Observational
Sponsor: The Society of Thoracic Surgeons (Other)
Collaborators: American College of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: TVTR-2012-01
Record Dates: First submitted 2012-11-14; First posted 2012-11-29 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2021-11

CONDITIONS: Aortic Valve Stenosis
Keywords: severe symptomatic native aortic valve stenosis; inoperable or high risk for open aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TAVR Patients: Will include all patients 18 years or over who undergo Transcatheter Aortic Valve Replacement (TAVR) for severe aortic stenosis. The sample size will include all patients entered into the Registry.
  Interventions: Procedure: Transcatheter Aortic Valve Replacement

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Replacement — Minimal invasive implantation of a biological prothesis in Aortic Position

SUMMARY:
The TVT Registry™ is a benchmarking tool developed to track patient safety and real-world outcomes related to the transcatheter aortic valve replacement (TAVR) procedure. Created by The Society of Thoracic Surgeons (STS) and the American College of Cardiology (ACC), the TVT Registry is designed to monitor the safety and efficacy of this new procedure for the treatment of aortic stenosis.

DETAILED DESCRIPTION:
Purpose of the Registry

The TVT Registry was designed to support a national surveillance system to assess the characteristics, treatments, and outcomes of patients receiving transcutaneous valve therapies. Patient-level data are submitted by participating hospitals to The Society of Thoracic Surgeons (STS) and American College of Cardiology Foundation's (ACCF) joint TVT Registry. The purposes of the TVT Registry include: (i) collecting pertinent and standardized data elements from participating hospitals, health care providers and others that measure and assess the quality of care for patients receiving TVT; (ii) providing confidential periodic reports to participating hospitals, health care providers and others, to evaluate and improve the quality of care in these areas; and (iii) permitting and fostering appropriate research based upon the data collected by means of the TVT Registry.

The secondary aim of the TVT Registry is to serve as a scalable data infrastructure for post market studies.

Background and Significance

Transcatheter valve therapies are now emerging into clinical practice from the research phase in the United States. The first of several approaches to replacing the aortic valve without open-chest surgery has now become a reality. Other valve and delivery systems are expected to be approved in the upcoming years. An Expert Consensus Document on Transcatheter Valve Therapy has outlined the initial technology, targeted patient population, and the multidisciplinary heart team and specialized facilities needed. The document also proposes the establishment of a national registry of patients with valvular heart disease that can collect and analyze data as these new valve treatment options become available. Surveillance of device performance, monitoring of long-term outcomes, and performance of comparative effectiveness research are some of the proposed uses of the registry.

Transcatheter valve therapies have emerged because of unmet patient needs. Furthermore, TVT has developed at a time when degenerative heart valve diseases of both the mitral and aortic valves are increasing in frequency as the population ages. With the introduction of the first TAVR commercial product, the targeted patient group is the "inoperable" patient who cannot receive the traditional therapy of surgical aortic valve replacement (SAVR). It is expected that TAVR will subsequently be extended to patients who have high risk with SAVR. The marked reduction of mortality by TAVR in the inoperable patients and the similar mortality of TAVR versus SAVR in the high risk patients provide patients with a new therapy with benefits but also with a different risk profile. Patients and their families will need to make informed decisions regarding the likelihood of having a mortality benefit, of improving their functional class and quality of life, of suffering a complication, and of choosing between different care options and therapeutic approaches.

For these patients there are unique issues such as the prioritization of the health related quality of life versus the quantity of life, the desire to preserve independence and avoid becoming a burden to families, and the need to clearly understand what about their current condition is reversible versus irreversible and linked to other conditions and aging. These issues become further highlighted when considering the considerable costs and other treatment burdens of the TVT technologies versus the disabling symptoms and recurrent hospitalizations caused by untreated severe valvular heart disease.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Transcatheter Aortic Valve Replacement must be furnished in a hospital with the appropriate infrastructre that includes, but is not limited to On site heart valve surgery program Cardiac catheterization lab or hybrid operating room with a fixed radiographic imaging system with flat panel fluoroscopy, offering quality imaging Non-invasive imaging such as echocardiography, vascular ultrasound, computed tomography and magnetic resonance Sufficient space, in a sterile environment, to accomodate necessary equipment for cases with and without complications Post-procedure intensive care facility with personnel experienced in managing patients who have undergone open-heart valve procedures Appropriate volume requirements
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2012-06 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-06 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | 30 day
  increase in the 30-day risk of adverse events among patients receiving TAVR

SECONDARY OUTCOMES:
Mortality | 1 year
  Proportion of patients who are alive with at least moderate functional improvement (defined as at least 10 point improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) from baseline) at 1 year after receiving TAVR

OTHER OUTCOMES:
Valve Academic Research Consortium (VARC) efficacy endpoint | 30 day
  30-day endpoints including mortality, stroke, stroke or transient ischemic attack (TIA), major vascular complications, valve related dysfunction requiring re-intervention, incident renal replacement therapy, life-threatening bleeding, and high-degree aortic valve (AV) block requiring permanent pacemaker implantation

CONTACTS AND LOCATIONS:
Overall Officials: John D Carroll, MD, Principal Investigator — American College of Cardiology; Fred H Edwards, MD, Principal Investigator — Society of Thoracic Surgeons
Locations (1):
- American College of Cardiology, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Tang GHL, Sengupta A, Alexis SL, Bapat VN, Adams DH, Sharma SK, Kini AS, Kodali SK, Ramlawi B, Gada H, Vora AN, Forrest JK, Kaple RK, Liu F, Reardon MJ. Outcomes of Prosthesis-Patient Mismatch Following Supra-Annular Transcatheter Aortic Valve Replacement: From the STS/ACC TVT Registry. JACC Cardiovasc Interv. 2021 May 10;14(9):964-976. doi: 10.1016/j.jcin.2021.03.040. PMID 33958170
- [Derived] Carroll JD, Mack MJ, Vemulapalli S, Herrmann HC, Gleason TG, Hanzel G, Deeb GM, Thourani VH, Cohen DJ, Desai N, Kirtane AJ, Fitzgerald S, Michaels J, Krohn C, Masoudi FA, Brindis RG, Bavaria JE. STS-ACC TVT Registry of Transcatheter Aortic Valve Replacement. Ann Thorac Surg. 2021 Feb;111(2):701-722. doi: 10.1016/j.athoracsur.2020.09.002. Epub 2020 Nov 16. PMID 33213826
- [Derived] Carroll JD, Mack MJ, Vemulapalli S, Herrmann HC, Gleason TG, Hanzel G, Deeb GM, Thourani VH, Cohen DJ, Desai N, Kirtane AJ, Fitzgerald S, Michaels J, Krohn C, Masoudi FA, Brindis RG, Bavaria JE. STS-ACC TVT Registry of Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2020 Nov 24;76(21):2492-2516. doi: 10.1016/j.jacc.2020.09.595. PMID 33213729
- [Derived] Attizzani GF, Patel SM, Dangas GD, Szeto WY, Sorajja P, Reardon MJ, Popma JJ, Kodali S, Chenoweth S, Costa MA. Comparison of Local Versus General Anesthesia Following Transfemoral Transcatheter Self-Expanding Aortic Valve Implantation (from the Transcatheter Valve Therapeutics Registry). Am J Cardiol. 2019 Feb 1;123(3):419-425. doi: 10.1016/j.amjcard.2018.10.041. Epub 2018 Nov 6. PMID 30527797
- [Derived] Abramowitz Y, Vemulapalli S, Chakravarty T, Li Z, Kapadia S, Holmes D, Matsouaka RA, Wang A, Cheng W, Forrester JS, Smalling R, Thourani V, Mack M, Leon M, Makkar RR. Clinical Impact of Diabetes Mellitus on Outcomes After Transcatheter Aortic Valve Replacement: Insights From the Society of Thoracic Surgeons/American College of Cardiology Transcatheter Valve Therapy Registry. Circ Cardiovasc Interv. 2017 Nov;10(11):e005417. doi: 10.1161/CIRCINTERVENTIONS.117.005417. PMID 29138245
- [Derived] Fanaroff AC, Manandhar P, Holmes DR, Cohen DJ, Harrison JK, Hughes GC, Thourani VH, Mack MJ, Sherwood MW, Jones WS, Vemulapalli S. Peripheral Artery Disease and Transcatheter Aortic Valve Replacement Outcomes: A Report From the Society of Thoracic Surgeons/American College of Cardiology Transcatheter Therapy Registry. Circ Cardiovasc Interv. 2017 Oct;10(10):e005456. doi: 10.1161/CIRCINTERVENTIONS.117.005456. PMID 29042398
- [Derived] Carroll JD, Vemulapalli S, Dai D, Matsouaka R, Blackstone E, Edwards F, Masoudi FA, Mack M, Peterson ED, Holmes D, Rumsfeld JS, Tuzcu EM, Grover F. Procedural Experience for Transcatheter Aortic Valve Replacement and Relation to Outcomes: The STS/ACC TVT Registry. J Am Coll Cardiol. 2017 Jul 4;70(1):29-41. doi: 10.1016/j.jacc.2017.04.056. PMID 28662805
- [Derived] Alfredsson J, Stebbins A, Brennan JM, Matsouaka R, Afilalo J, Peterson ED, Vemulapalli S, Rumsfeld JS, Shahian D, Mack MJ, Alexander KP. Gait Speed Predicts 30-Day Mortality After Transcatheter Aortic Valve Replacement: Results From the Society of Thoracic Surgeons/American College of Cardiology Transcatheter Valve Therapy Registry. Circulation. 2016 Apr 5;133(14):1351-9. doi: 10.1161/CIRCULATIONAHA.115.020279. Epub 2016 Feb 26. PMID 26920495
- [Derived] Mack MJ, Brennan JM, Brindis R, Carroll J, Edwards F, Grover F, Shahian D, Tuzcu EM, Peterson ED, Rumsfeld JS, Hewitt K, Shewan C, Michaels J, Christensen B, Christian A, O'Brien S, Holmes D; STS/ACC TVT Registry. Outcomes following transcatheter aortic valve replacement in the United States. JAMA. 2013 Nov 20;310(19):2069-77. doi: 10.1001/jama.2013.282043. PMID 24240934
- [Derived] Carroll JD, Edwards FH, Marinac-Dabic D, Brindis RG, Grover FL, Peterson ED, Tuzcu EM, Shahian DM, Rumsfeld JS, Shewan CM, Hewitt K, Holmes DR Jr, Mack MJ. The STS-ACC transcatheter valve therapy national registry: a new partnership and infrastructure for the introduction and surveillance of medical devices and therapies. J Am Coll Cardiol. 2013 Sep 10;62(11):1026-34. doi: 10.1016/j.jacc.2013.03.060. Epub 2013 May 1. PMID 23644082
- See also: Link to homepage for STS/ACC TVT Registry — https://www.ncdr.com/TVT/Home/Default.aspx